CLINICAL TRIAL: NCT03296618
Title: Phase I Clinical Study of Intracerebral Transplantation of Neural Stem Cells for the Treatment of Ischemic Stroke
Brief Title: Intracerebral Transplantation of Neural Stem Cells for the Treatment of Ischemic Stroke
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suzhou Neuralstem Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Neuralstem Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS2012-1
Record Dates: First submitted 2017-09-22; First posted 2017-09-28 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Ischemic Motor Stroke, Chronic
Keywords: chronic stroke; neural stem cell; transplant; paralysis
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NSI-566 neural stem cell implantation (Experimental)
  Interventions: Drug: NSI-566

INTERVENTIONS:
Drug: NSI-566 — Dosing will consist of a one-time stereotactic, intracranial injection of a hNSC line, NSI-566, ranging from 1.2×107 cells to 8×107 cells, as tolerated.

SUMMARY:
The study is to determine the safety of human neural stem cell transplantation for the treatment of paralysis and related symptoms due to chronic motor stroke and to determine the maximum tolerated dose.

DETAILED DESCRIPTION:
This is a Phase I study of human neural stem cell transplantation for the treatment of chronic motor stroke. This single-site, Phase I, open-label study may enroll up to 18 patients across 5 cohorts of ascending doses of human neural stem cells to define maximal tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the requirements of the study, provide written informed consent, understand and provide written authorization for the use and disclosure of Protected Health Information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) Privacy Ruling] and comply with the study procedures
2. Men and women 30-65 years old
3. Women must have a negative serum pregnancy test and practice an acceptable method of contraception or be of non-childbearing potential (post-menopausal for at least 2 years or who have undergone hysterectomy or oophorectomy or surgical sterilization)
4. At least 3 months but no more than 24 months from time of stroke, with a motor neurological deficit
5. Documented history of completed ischemic stroke in subcortical region of MCA or lenticulostriate artery with or without cortical involvement, with correlated findings by MRI
6. Modified Rankin Score of 2, 3 or 4
7. FMMS score of 55 or less;
8. Two evaluations at approximately 3 weeks apart prior to surgery with less than +/- 4 point change in the NIHSS
9. Able and willing to meet all follow-up requirements
10. Able and willing to undergo post-physical therapy/rehabilitation

Exclusion Criteria:

1. Any disabling psychological or psychiatric disorders which may confound the study
2. History of more than one symptomatic stroke, TIAs allowed
3. History of another major neurological disease or injury
4. Cerebral infarct size >8cm in any one measurement
5. Myocardial infarction within the prior 3 months
6. History of seizures or current use of antiepileptic medication
7. Receipt of any investigational drug or device within 30 days
8. Receipt of any cell infusion other than blood transfusion
9. Any concomitant medical disease or condition noted below:

   1. Coagulopathy with INR > 1.4 at the time of surgery
   2. Panel Reactive Antibodies (PRA) > 20% at initial screen
   3. Active infection at the time of surgery
   4. Active hypotension requiring vasopressor therapy
   5. Skin breakdown over the site of surgery
   6. Active or history of malignancy
   7. Primary or secondary immune deficiency
   8. Persistent MRI artifact that would prevent imaging pre and post-operation or unable to undergo MRI
   9. Creatinine >115μmol/L, liver function tests (SGOT/SGPT, Bilirubin, Alk Phos) > 2x upper limit of normal, hematocrit/hemoglobin < 30/10, total WBC < 4000/mm3,platelet count <100,000/mm3, uncontrolled hypertension (systolic > 180mmHg or diastolic> 100mmHg) or uncontrolled diabetes (defined as hemoglobin A1C>8%), evidence of GI bleeding by hemoccult test,positive tuberculosis (TB test: PPD/Mantoux), hepatitis B or C, or human immunodeficiency virus (HIV)
10. Presence of any of the following conditions:

    1. Current drug abuse or alcoholism
    2. Unstable medical conditions
    3. Unstable psychiatric illness including psychosis and untreated major depression
11. Any condition that the Investigator or primary physician feels may interfere with participation in the study or may endanger the subject
12. Any condition that the surgeon feels may pose complications for the surgery
13. Known hypersensitivity to tacrolimus or methylprednisolone
14. Unable or unwilling to participate in physical and/or occupational therapy or return to clinic for follow up examinations as scheduled
15. Inability to provide informed consent as determined by screening protocol.
16. Use of antiplatelet drugs less than 2 weeks before surgery

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2012-06; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 24 months

SECONDARY OUTCOMES:
Clinical improvement using NIH Stroke Scale | 12 months
Clinical improvement using Modified Rankin Scale | 12 months
Clinical improvement using Fugl-Meyer Motor Score | 12 months
Clinical Improvement using Mini-mental State Examination | 12 months

OTHER OUTCOMES:
MRI analysis of transplant site | 12 months
PET analysis of transplant site | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xu Ruxiang, M.D, Principal Investigator — BaYi Brain Hospital, Army General Hospital
Locations (1):
- Ba Yi Brain Hospital, Beijing, China

REFERENCES:
- [Background] Glass JD, Boulis NM, Johe K, Rutkove SB, Federici T, Polak M, Kelly C, Feldman EL. Lumbar intraspinal injection of neural stem cells in patients with amyotrophic lateral sclerosis: results of a phase I trial in 12 patients. Stem Cells. 2012 Jun;30(6):1144-51. doi: 10.1002/stem.1079. PMID 22415942
- [Background] Boulis NM, Federici T, Glass JD, Lunn JS, Sakowski SA, Feldman EL. Translational stem cell therapy for amyotrophic lateral sclerosis. Nat Rev Neurol. 2011 Dec 13;8(3):172-6. doi: 10.1038/nrneurol.2011.191. PMID 22158518
- [Background] Lunn JS, Sakowski SA, Hur J, Feldman EL. Stem cell technology for neurodegenerative diseases. Ann Neurol. 2011 Sep;70(3):353-61. doi: 10.1002/ana.22487. PMID 21905078
- [Background] Lunn JS, Sakowski SA, Federici T, Glass JD, Boulis NM, Feldman EL. Stem cell technology for the study and treatment of motor neuron diseases. Regen Med. 2011 Mar;6(2):201-13. doi: 10.2217/rme.11.6. PMID 21391854